CLINICAL TRIAL: NCT00154505
Title: Effects of Lateral Trunk Support on Spinal Alignment in Spinal Cord Injured Persons
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9261701245; NSC 91-2314-B-002-393; NSC 92-2314-B-002-084
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2002-08

CONDITIONS: Scoliosis; Spinal Cord Injury
Keywords: Scoliosis; Spinal Cord Injury; Lateral Trunk Support; Radiography
MeSH Terms: conditions — Scoliosis; Spinal Cord Injuries

INTERVENTIONS:
Device: Lateral trunk support of wheelchair seating

SUMMARY:
The effects of lateral trunk supports (LTS) in special seating on the spinal alignment of 17 spinal cord injured (SCI) subjects with scoliosis were studied using bi-planar radiographs. The LTS improved significantly the functional scoliotic spinal alignment in the frontal and sagittal planes regardless of the severity of scoliosis.

DETAILED DESCRIPTION:
SCI patients often develop progressive scoliosis due to loss of muscular support to maintain good sitting posture. Special seating with LTS has been widely used in clinical practice to improve their sitting postures. However, little is known as to how this can affect the scoliotic curve.The purpose of this study was to investigate the effects of lateral trunk supports (LTS) in special seating on the spinal alignment of spinal cord injured (SCI) individuals with scoliosis.

Ten male and seven female SCI subjects with scoliosis sat on an experimental chair with and without LTS while radiographs of the spine in the anteroposterior and lateral directions were taken. Radiographs of the spine in the A-P and lateral directions were taken with a digital radiographic imaging system (Saturn 9000 M, Comed., Korea). For each direction, the complete image of the spine was obtained from separate x-ray images of the upper and lower trunk due to the limited field of view of the x-ray machine. The Cobb angles and scoliotic indices based on the anteroposterior radiographic images and the angles of the thoracic and lumber spine based on lateral were calculated.

ELIGIBILITY:
Inclusion Criteria:

* (1) C4-T12 SCI, (2) onset over 1 year, (3) sitting on the wheelchair more than 4 hours per day, (4) diagnosed thoracic or lumbar scoliosis through A-P radiographs, (5) flexible scoliosis, confirmed by supine and side-lying bending radiographs.

Exclusion Criteria:

* inflexible scoliosis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2002-09; Study Completion 2004-11

PRIMARY OUTCOMES:
Spinal aligamnet(Cobb angle)

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Fen Mao, MS, Principal Investigator — National Taiwan University
Locations (1):
- School of Occupational Therapy, National Taiwan University, Taipei, Taiwan